CLINICAL TRIAL: NCT03290924
Title: Accelerating Newborn Survival in Ghana Through a Low-dose, High-frequency Health Worker Training Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jhpiego (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: OPP1087303
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Stillbirth; Neonatal Death
Keywords: institutional delivery
MeSH Terms: conditions — Stillbirth; Perinatal Death

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Low-dose high-frequency health worker training approach to update skilled birth attendants in key evidence-based intrapartum and immediate newborn care practices
  Interventions: Behavioral: Low dose high frequency health worker training approach
- Comparison (Active Comparator): Training on data collection and reporting
  Interventions: Behavioral: Active Comparison

INTERVENTIONS:
Behavioral: Low dose high frequency health worker training approach — * Two 4-day training sessions for skilled birth attendants
  * 1-day peer practice coordinator training after first training session
  * Weekly, peer-led practice sessions using MamaNatalie® and NeoNatalie™ anatomic models
  * SMS reminder messages and quizzes
  * Routine telephone calls between master mentors and peer practice coordinators, and between project staff and master mentors
  * Health information officer training
  * Data collection and use training
  * Supply of simulators, newborn resuscitation equipment, and delivery sets
  Arms: Intervention
Behavioral: Active Comparison — Training on data collection and reporting
  Arms: Comparison

SUMMARY:
This study assesses the effect of a low-dose, high-frequency training approach on long-term evidence-based skill retention among skilled birth attendants and impact on adverse birth outcomes at hospitals in Ghana.

DETAILED DESCRIPTION:
In-service training for skilled birth attendants (SBAs) is one of the most common interventions to address lack of knowledge and skills. However, these training interventions are seldom evaluated for effectiveness in improving learning or performance.

This study study is a cluster-randomized waitlist trial implemented in 40 public and mission hospitals in Ghana. It assesses the effect of a low-dose, high-frequency (LDHF) training approach to update hospital-based SBAs in key evidence-based intrapartum and immediate newborn care practices, using current global guidelines.The LDHF approach includes two 4-day onsite sessions (low dose) with weekly practice sessions, SMS quizzes and reminders, and mentoring via mobile phone and onsite visits between trainings (high frequency). The low-dose sessions include competency acquisition through simulation, case-based learning, and small content packages spread over short time intervals.

Eligible hospitals will be stratified by geographic region and caseload, and then randomly assigned to one of four implementation waves. The pipeline randomization allows for rigorous evaluation while the program is rolled out to all facilities.

ELIGIBILITY:
INCLUSION CRITERIA - FACILITIES:

* Public or faith based hospital
* At least three skilled birth attendants on staff
* At least 30 births per month

EXCLUSION CRITERIA - FACILITIES:

* Private hospital
* Public or faith based hospital with less than three skilled birth attendants on staff
* Public or faith based hospital with less than 30 births per month

INCLUSION CRITERIA - SERVICE PROVIDERS:

* Health providers who attend births in participating health facilities and consent to be assessed at the time of enrollment and at several points in time over the study period

EXCLUSION CRITERIA - SERVICE PROVIDERS:

* Health providers who decline to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
institutional twenty-four hour newborn mortality rate | 1 day
  death within 24 hours, or before discharge, of a newborn who breathed at birth
institutional intrapartum stillbirth rate | 1 day
  proportion of all facility births that resulted in intrapartum stillbirth

SECONDARY OUTCOMES:
skilled birth attendant knowledge and skills | Pre-test (before training) - post-test (immediately after training) - endline (12 months)
  score on written and practical examinations on routine and emergency obstetric and newborn care

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Gomez, Principal Investigator — Senior Technical Advisor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gomez PP, Nelson AR, Asiedu A, Addo E, Agbodza D, Allen C, Appiagyei M, Bannerman C, Darko P, Duodu J, Effah F, Tappis H. Accelerating newborn survival in Ghana through a low-dose, high-frequency health worker training approach: a cluster randomized trial. BMC Pregnancy Childbirth. 2018 Mar 22;18(1):72. doi: 10.1186/s12884-018-1705-5. PMID 29566659